CLINICAL TRIAL: NCT01723215
Title: Prevention of Posttraumatic Symptoms in IDF Soldiers Using Attention Bias Modification (ABM): A Randomized Controlled Trial
Brief Title: Prevention of Combat-related PTSD Using Attention Bias Modification (ABM): A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: Medical Corps, Israel Defense Force (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TelAvivU
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: PTSD
Keywords: Attention bias modification; resilience; combat; PTSD; Depression; Anxiety
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active ABMT8 (Active Comparator): Active ABMT8 8 active ABMT sessions (10 min. each, over 7-8 weeks) designed to promote adaptive threat attendance
  Interventions: Behavioral: Active ABMT8
- Active ABMT4 (Active Comparator): Active ABMT4 4 active ABMT sessions (10 min. each, over 7-8 weeks) designed to promote adaptive threat attendance
  Interventions: Behavioral: Active ABMT4
- Control (No Intervention): Control: will not receive any intervention
- Placebo (Placebo Comparator): Placebo: will receive 4 training sessions(10 min. each, over 7-8 weeks) using the same task and stimuli as in the active arms, but not designed to change attention patterns
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Active ABMT8 — Active ABMT8 8 active ABMT sessions (10 min. each, over 7-8 weeks) designed to promote adaptive threat attendance
  Arms: Active ABMT8
Behavioral: Active ABMT4 — Active ABMT4 4 active ABMT sessions (10 min. each, over 7-8 weeks) designed to promote adaptive threat attendance
  Arms: Active ABMT4
Behavioral: Placebo — Placebo: will receive 4 training sessions(10 min. each, over 7-8 weeks) using the same task and stimuli as in the active arms, but not designed to change attention patterns
  Arms: Placebo

SUMMARY:
Military deployment to combat zones involves exposure to trauma at a higher than average rate and therefore presents a unique opportunity to study predisposing factors to posttraumatic stress reactions and test strategies designed to prevent and ameliorate posttraumatic symptoms. Decades of scientific research on the origins of resilience and vulnerability to combat-related posttraumatic stress symptoms revealed various predisposing and protective factors. All these factors however, offer limited opportunity for systematic pre-deployment prevention efforts. Considering the magnitude of psychological adjustment difficulties encountered by combat personnel in deployment and the limited access to existing evidence-based therapies for PTSD, the development and testing of a novel evidence-based and theory-driven prevention protocol for these problems is of considerable significance. The current study translates cognitive-neuroscience knowledge and attention bias modification research into a novel computerized training tool that could be easily delivered to soldiers during different stages of the deployment cycle. If proved efficacious in reducing risk for posttraumatic symptoms ABMT could be integrated into the Army's resilience training program. Thus, we propose a longitudinal double-blind randomized controlled study of ABMT in soldiers. We will assess attention bias and symptoms before deployment, will randomly assign soldiers to either 8 ABMT sessions, 4 ABMT sessions, 8 Placebo training sessions, or no training. Following 6 months of deployment to combat zone symptoms will be assessed again.

ELIGIBILITY:
Inclusion Criteria:

* combat soldiers

Exclusion Criteria:

* Fluent Hebrew

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 862 (Actual)
Dates: Start 2012-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Changes in PTSD symptoms(PCL) | Pre-treatment(baseline), after first deployment, 10 days after combat, 4 months after combat
  1. pre-treatment 2.after first deployment 3.10 days after combat 4. 4 months after combat
Probable PTSD diagnosis(CAPS) | Four months after combat
  Four months after combat

SECONDARY OUTCOMES:
Changes in Depression(PHQ-9)) and Anxiety(STAI) | Pre-treatment(baseline), after first deployment, 10 days after combat, 4 months after combat
  1. Pre-treatment(baseline) 2.after first deployment 3.10 days after combat 4. 4 months after combat

OTHER OUTCOMES:
Attention Bias Scores | Pre-traetment baseline and in deployment
  Attention bias scores measured in milliseconds using the dot-probe task

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University; Eyal Fruchter, Principal Investigator — Mental Health Department IDF
Locations (1):
- IDF Military camps, Beersheba, Israel

REFERENCES:
- [Background] Bar-Haim Y. Research review: Attention bias modification (ABM): a novel treatment for anxiety disorders. J Child Psychol Psychiatry. 2010 Aug;51(8):859-70. doi: 10.1111/j.1469-7610.2010.02251.x. Epub 2010 May 6. PMID 20456540
- [Background] Bar-Haim Y, Holoshitz Y, Eldar S, Frenkel TI, Muller D, Charney DS, Pine DS, Fox NA, Wald I. Life-threatening danger and suppression of attention bias to threat. Am J Psychiatry. 2010 Jun;167(6):694-8. doi: 10.1176/appi.ajp.2009.09070956. Epub 2010 Apr 15. PMID 20395400
- [Derived] Wald I, Fruchter E, Ginat K, Stolin E, Dagan D, Bliese PD, Quartana PJ, Sipos ML, Pine DS, Bar-Haim Y. Selective prevention of combat-related post-traumatic stress disorder using attention bias modification training: a randomized controlled trial. Psychol Med. 2016 Sep;46(12):2627-36. doi: 10.1017/S0033291716000945. Epub 2016 Jul 5. PMID 27377418